CLINICAL TRIAL: NCT05500885
Title: The Clinical Effectiveness of Pulsed Electromagnetic Field Therapy on the Management of Chronic Ankle Instability: A Double-Blinded Randomized Controlled Trial
Brief Title: The Clinical Effectiveness of Pulsed Electromagnetic Field Therapy on the Management of Chronic Ankle Instability
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022.263-T
Record Dates: First submitted 2022-07-27; First posted 2022-08-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Chronic Ankle Instability
MeSH Terms: interventions — carboxyamido-triazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active PEMF therapy for chronic ankle instability (Experimental): Participants will be randomized into 1:1 allocation, blocked randomization with 20 participants in the PEMF group and 20 participants in the sham group. Each allocation will be assigned with a unique RFID (generated during block randomization by the PEMF supplier service) recognizable by the PEMF machine.
  Interventions: Device: PEMF device, Quantum Tx, Singapore
- Sham PEMF therapy for chronic ankle instability (Sham Comparator): Control group will receive sham treatment on top of a standard rehabilitation (muscle strengthening and balance training).
  Interventions: Other: Standard rehabilitation and sham PEMF therapy for CAI

INTERVENTIONS:
Device: PEMF device, Quantum Tx, Singapore — The options of the appliance will be adjusted to 1.5mT, 10Hz on the diseased leg for 10 minutes.
  Arms: Active PEMF therapy for chronic ankle instability
Other: Standard rehabilitation and sham PEMF therapy for CAI — Balance training and muscle strengthening
  Arms: Sham PEMF therapy for chronic ankle instability

SUMMARY:
This study aims to investigate the clinical effectiveness of PEMF as an adjunct to a program of standard rehabilitation for the treatment of chronic ankle instability. The study objective is to establish whether PEMF plus standard rehabilitation in people with chronic ankle instability compared to standard rehabilitation. This study also investigates the effects of PEMF on pain, functional outcomes, and mechanical and morphological properties of peroneal muscles in chronic ankle instability. Investigators hypothesize that pulsed electromagnetic field therapy is effective in reducing pain, improving functional outcomes, and restoring mechanical and morphological properties.

This study is a double-blinded, randomized controlled trial to investigate the clinical effects of pulsed electromagnetic field therapy (PEMF) for chronic ankle instability. Participants will be recruited from the outpatient clinic of the orthopedic and traumatology department at Prince of Wales Hospital.

40 patients aged between 18 to 60 years old with CAI will be invited to join this trial after informed consent. Participants will be randomized to any of the 2 groups: the intervention group (n=20; PEMF (Quantum Tx) treatment), and the control group (n=20; sham treatment with dummy exposure to PEMF).

For Chronic Ankle Instability patients: baseline measurements of all self-reported outcomes, functional outcomes, and ultrasound imaging assessments, such as dynamic balance, static balance, single leg hop test, gait evaluation, dorsiflexion range of motion, and eversion muscle strength.

DETAILED DESCRIPTION:
The primary objective is to investigate the effectiveness of PEMF therapy on the clinical and functional outcomes in the CAI population. We hypothesize that PEMF therapy will effectively improve the clinical and functional outcomes of patients with CAI.

Methods: This is a prospective, randomized, double-blinded, placebo-controlled trial with blinded assessors. A total of 40 adults with CAI will be recruited and randomly allocated into either the intervention or control group. In the intervention group, the participants (n=20) will receive active PEMF therapy and standard exercise training, while the control group (n=20) will receive sham-PEMF therapy and standard exercise training. The PEMF intervention will last for 8 weeks. The primary and secondary outcomes will be evaluated at baseline, week 4, week 8, 3rd month, 6th month after the PEMF therapy.

Rationale: Pulse electromagnetic field therapy (PEMF) as an adjunct biophysical therapy can improve stability by mitigating peroneal muscle weakness and activating peroneal muscle. Therefore, we postulate the combination of standard care (muscle strengthening, balance training, and range of motion exercise) augmented with pulse electromagnetic field therapy elicits a significant improvement in postural control stability and peroneal muscle weakness.

ELIGIBILITY:
* Inclusion in the CAI stratum:
* Requires a history of at least one significant sprain > 12 months prior to consent
* Continued perceived or episodic "giving way" of the ankle
* Reported Cumberland Ankle Instability Tool (CAIT score < 24)

Exclusion Criteria for CAI:

* A history of surgeries or fractures of either lower extremity limbs
* Concomitant lower extremity pathology, e.g. vascular disease and osteoarthritis
* Inadequate muscle strength in lower limb which require ambulation support (e.g., crutches) or any vestibular or balance disorders
* Pregnancy
* Cognitive impairment/Neurological conditions, and neurological disorders (e.g. dementia) -Concussion within the last 6 months
* Bilateral instability condition
* Regular use of medicine or antibiotics
* Metal implantation in their body
* Unable to walk at enrolment
* Non-removable cast

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Centre of pressure during single leg stance for chronic ankle instability | Baseline to 6 months
  Static balance will be conducted in double-leg and single leg stance with eyes opened and closed on the Tekscan pressure mat.

SECONDARY OUTCOMES:
Y balance test for chronic ankle instability | Baseline to 6 months
  Dynamic balance
Dorsiflexion Range of motion for chronic ankle instability | Baseline to 6 months
  The range of motion (ROM) will be measured by weight bearing lunge test (WBLT).
Foot muscle strength for chronic ankle instability population | Baseline to 6 months
  Foot muscle strength will be carried out using a handheld dynamometer during ankle dorsiflexion, plantar flexion, inversion and eversion.
Ultrasound imaging for peroneal muscle in chronic ankle instability patients | Baseline to 6 months
  The ultrasound imaging assessment of the peroneal muscle will be performed using Aixplorer (Supersonic Imagine, Aix-en-Provence, France).
Short Form 36 questionnaire (SF-36) | Baseline to 6 months
  The 36 questions on the SF-36 are meant to reflect 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social function, emotional role, and mental health. The categories of physical role and emotional role reflect performance at the activity and participation levels. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
CAIT score | Baseline to 6 months
  Cumberland Ankle Instability Tool (CAIT) score is a valid and reliable 9-item instrument used to identify self-perceived ankle instability. The instrument is scored on a 0 (worst) to 30 (best) scale, where a cut-off point of ≤ 24 denotes the presence of instability.
Lateral step-down test (LSDT) | Baseline to 6 months
  LSDT is a clinical measurement that evaluates dynamic postural stability deficits and potential lower extremity injury. It measures the coordination of the lower limb joints, neuromuscular control, strength, pelvic stability, and range of motion.
The Manchester-Oxford Foot Questionnaire (MOxFQ) | Baseline to 6 months
  It is validated 16-item, patient-reported outcome measure of foot and ankle pain and function
Numerical pain scale for chronic ankle instability | Baseline to 6 months
  The numerical pain scale requires participants to rate their pain on a defined scale from 0-100. 0 refers to no pain while 100 refers to severe pain. Lower scores mean a better outcome.
Foot and ankle measure | Baseline to 6 months
  Foot and Ankle Ability Measure (FAAM) will be used to assess the foot and ankle functional limitations among CAI individuals.
Dorsiflexion range of motion | Baseline to 6 months
  Weight-bearing lung test (WBLT), based on the knee-to-wall principle, is a valid and reliable assessment that measures the dorsiflexion range of motion in CAI population.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chia CSM, Fu SC, He X, Cheng YY, Franco-Obregon A, Hua Y, Yung PS, Ling SK. The clinical effects of pulsed electromagnetic field therapy for the management of chronic ankle instability: a study protocol for a double-blind randomized controlled trial. Trials. 2024 Dec 3;25(1):808. doi: 10.1186/s13063-024-08639-z. PMID 39627831